CLINICAL TRIAL: NCT01068327
Title: A Phase 1 Study of Hypofractionated Stereotactic Radiotherapy and Concurrent HIV Protease Inhibitor Nelfinavir as Part of a Neoadjuvant Regimen in Patients With Locally Advanced Pancreatic Cancer
Brief Title: Stereotactic Radiation, Nelfinavir Mesylate & Neoadjuvant Chemotherapy in Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0441-07-FB; NCI-2009-01443 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA036727 (NIH); NCT00705393 (obsolete NCT alias)
Record Dates: First submitted 2010-01-25; First posted 2010-02-12 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Adenocarcinoma of the Pancreas; Stage III Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Leucovorin; Fluorouracil; Nelfinavir; Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (SRT, radiosensitizer, and chemotherapy) (Experimental): See Detailed Description
  Interventions: Drug: gemcitabine hydrochloride; Drug: leucovorin calcium; Drug: fluorouracil; Drug: nelfinavir mesylate; Radiation: stereotactic body radiation therapy; Radiation: hypofractionated radiation therapy; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Drug: nelfinavir mesylate — Given PO
  Other Names: Viracept
Radiation: stereotactic body radiation therapy — Undergo radiotherapy
  Other Names: SBRT; stereotactic radiation therapy; stereotactic radiotherapy
Radiation: hypofractionated radiation therapy — Undergo radiotherapy
Procedure: therapeutic conventional surgery — Undergo surgery

SUMMARY:
This phase I trial is studying the side effects and best dose of stereotactic radiation therapy and nelfinavir mesylate when given together with gemcitabine hydrochloride, leucovorin calcium, and fluorouracil in treating patients with locally advanced pancreatic cancer. Stereotactic radiation therapy may be able to send x-rays directly to the tumor and cause less damage to normal tissue. Drugs, such as nelfinavir mesylate, may make tumor cells more sensitive to radiation therapy. Drugs used in chemotherapy, such as gemcitabine hydrochloride, leucovorin calcium, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving stereotactic radiation therapy and nelfinavir mesylate together with combination chemotherapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the safety, dose-limiting toxicities and maximally tolerated dose of hypofractionated stereotactic radiotherapy concurrently with nelfinavir in patients with locally advanced pancreatic cancer given as part of a neoadjuvant chemoradiation therapy regimen.

SECONDARY OBJECTIVES:

I. To evaluate the surgical complete resection rate. II. To evaluate the pathological response. III. To evaluate tumor response on computed tomography (CT)/magnetic resonance imaging (MRI).

IV. To evaluate the correlation between the radiologic response and pathologic response.

TERTIARY OBJECTIVES:

I. To measure phospho-AKT expression in pancreatic tumor tissue prior to and following the neoadjuvant chemo-radiation program. (Correlative) II. To measure nelfinavir pharmacokinetics at steady-state. (Correlative) III. To measure the pharmacogenomic status of CYP2C19*2 (G681A) in the study population. (Correlative)

OUTLINE: This is a dose-escalation study of stereotactic radiotherapy (SRT) and concurrent nelfinavir mesylate.

NEOADJUVANT THERAPY: Patients receive gemcitabine hydrochloride intravenously (IV) over 30 minutes, leucovorin calcium IV over 30 minutes, and fluorouracil IV continuously over 24 hours on days 1 and 8. Treatment repeats every 3 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity. Patients then receive nelfinavir mesylate orally (PO) twice daily (BID) beginning in week 9 and continuing until the completion of SRT or until 14 days after the completion of SRT. Patients undergo concurrent SRT once daily for 5 days in week 11.

SURGERY AND ADJUVANT CHEMOTHERAPY: Approximately 2-3 weeks after completion of SRT, patients undergo restaging to evaluate disease response. Patients with resectable or potentially resectable disease and no metastasis undergo definitive surgery 2-3 weeks later. Approximately 1 month after surgery, these patients receive three additional courses of gemcitabine hydrochloride, leucovorin calcium, and fluorouracil as above. Patients with unresectable disease that is stable or responsive at the time of surgical exploration may resume treatment with gemcitabine hydrochloride, leucovorin calcium, and fluorouracil as above in the absence of disease progression or unacceptable toxicity. Patients with metastatic disease at the time of restaging are removed from the study.

After completion of study treatment, patients are followed every 3 months for 1 year, every 4 months for 1 year, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* The time between other investigational agents and enrollment on this study is at least 30 days
* Pathologically confirmed adenocarcinoma of the pancreas
* Patients have localized or locally advanced disease with no evidence of distant metastases
* The maximum dimension of the tumor must be =< 8 cm
* Karnofsky Performance Status of 60% or better
* Patients with biliary or gastroduodenal obstruction must have drainage or surgical bypass prior to starting chemoradiation
* Patients who received chemotherapy > 5 years ago for malignancies other than pancreatic cancer are eligible, provided that chemotherapy was completed > 5 years ago and that there is no evidence of the second malignancy at the time of study entry
* Patients who received radiation therapy > 5 years ago for malignancies other than pancreatic cancer and whose radiation therapy field is not overlapping with the 20% isodose line of current radiation field are eligible, provided that radiation therapy was completed > 5 years ago and that there is no evidence of the second malignancy at the time of study entry
* All malignant disease must be able to be encompassed within a single irradiation field
* All patients must have radiographically assessable disease
* Patients must have a absolute granulocyte count (AGC) greater than or equal to 1500/uL and platelet count greater than or equal to 100,000/uL
* Patients must have a serum creatinine less than or equal to 2 mg/dL and total bilirubin less than or equal to 2.0 mg/dL in the absence of biliary obstruction
* If the patient has biliary obstruction, biliary decompression will be required; either endoscopic placement of biliary stent (7 French or greater) or percutaneous transhepatic drainage are acceptable; once biliary drainage has been established, institution of gemcitabine therapy may proceed when the total bilirubin falls to below 4.0 mg/dL
* The patient must be aware of the neoplastic nature of his/her disease and willingly provide written, informed consent after being informed of the procedure to be followed, the experimental nature of the therapy, alternatives, potential benefits, side-effects, risks, and discomforts
* Patients may have had prior chemotherapy for pancreatic cancer
* Any prior therapy is acceptable except radiation to the abdomen

Exclusion Criteria:

* Patients receiving the following drugs will be clinically evaluated as to whether dosage/medication can be changed to permit patient on study: carbamazepine; phenobarbital; phenytoin; rifabutin; sildenafil; atorvastatin; cyclosporine; tacrolimus; sirolimus; methadone; ethinyl estradiol; azithromycin
* Patients who can not undergo staging laparoscopy and marker implantation; this may include patients with a prior history of multiple abdominal operations in which laparoscopy may not be technically feasible or potentially harmful
* The patient is eligible if they have a common bile duct stent adjacent to the tumor that may be used as an internal marker, or if the patient has already had a staging laparoscopy without marker implantation and the markers can be implanted (by interventional radiology) prior to the beginning of radiation therapy
* History of allergy to chemotherapy agents or to antiemetics appropriate for administration in conjunction with protocol-directed chemotherapy
* Uncontrolled inter-current illness including, but not limited to ongoing or active infection requiring intravenous antibiotics, symptomatic congestive heart failure, unstable angina pectoris, or serious, uncontrolled cardiac arrhythmia, that might jeopardize the ability of the patient to receive the chemotherapy program outlined in this protocol with reasonable safety
* Patients with human immunodeficiency virus (HIV) infection, or hepatic insufficiency
* Patients may not be receiving or have received any other investigational agents during/or within 1 month prior to treatment with NFV (nelfinavir mesylate)
* Patients who can not take oral medications
* Patients with active duodenal ulcer or bleeding or history of a gastrointestinal fistula or perforation or other significant bowel problems (severe nausea, vomiting, inflammatory bowel disease and significant bowel resection)
* Patients with prior malignancy will be excluded EXCEPT for adequately treated basal cell or squamous cell skin cancer, adequately treated noninvasive carcinomas, or other cancers from which the patient has been disease-free for at least 5 years
* Patients receiving the following drugs that are contraindicated with NFV will be excluded: amiodarone; quinidine; rifampin; dihydroergotamine; ergonovine; ergotamine; methylergonovine; St. John's wort (hypericum perforatum); lovastatin; simvastatin; pimozide; midazolam; triazolam
* Pregnant and nursing women are excluded from this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2007-11-05; Primary Completion 2013-08-01 (Actual); Study Completion 2015-02-01 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity as assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v3.0 | Within 1 month of surgery
  Due to delayed toxicities attributable to radiotherapy, all toxicities observed within 1 month of surgery will be scored. Toxicity will be graded and tabled by dose levels.
Maximally tolerated dose (MTD) of stereotactic radiotherapy and concurrent nelfinavir mesylate | 3 patients will initially be treated at each dose level (4 levels); a minimum of 1 month of observation after surgery is required in all 3 patients before escalation
  The MTD of SRT/nelfinavir mesylate is defined as the highest dose level at which no greater than one dose-limiting toxicity is observed in 6 patients.

SECONDARY OUTCOMES:
Rate of complete surgical resection | At the time of surgery (2-3 weeks after completion of SRT)
  At the MTD, the rate of surgical complete resection with 90% exact binomial confidence intervals will be calculated.
Pathological response | Pre- to post-treatment
  At the MTD, the rate of pathologic response with 90% exact binomial confidence intervals will be calculated.
Tumor response on CT/MRI | Change from pre- to post-treatment
  Pre- to post-treatment changes in tumor size on CT or MRI scan (if CT is not sufficient).
Radiologic response and pathologic response | Pre- to post-treatment
  Correlation between the radiologic response and pathologic response
Phospho-AKT expression in pancreatic tumor tissue (correlative) | Pre- to post-nelfinavir mesylate
  Exploratory analyses will compare pre- to post-nelfinavir mesylate treatment changes in Akt levels between patients who achieve or do not achieve R0 resection by the nonparametric Wilcoxon rank sum test.
Pharmacokinetics of nelfinavir mesylate (correlative) | After at least 1 week of NFV: *0 h (trough); *After NFV dosing: 1, 2, 3, 4, 5, 6, 8, and 12 h
  The data will be modeled using WinNonLin Pro version 4.1. The pharmacokinetic parameters will be presented as the mean and standard deviation.
Pharmacogenomic status of CYP2C19*2 (G681A) (correlative) | Enrollment, at the time of planned tumor tissue procurement, and at the time that re-staging studies are done
  There is currently insufficient clinical data to indicate whether any of the specific polymorphisms proposed to be studied, particularly those subjects with a heterozygous state, will correlate with meaningful differences in the pharmacokinetic parameters of nelfinavir mesylate. These analyses must therefore be exploratory in nature.

CONTACTS AND LOCATIONS:
Overall Officials: Chi Lin, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Derived] Lin C, Verma V, Ly QP, Lazenby A, Sasson A, Schwarz JK, Meza JL, Are C, Li S, Wang S, Hahn SM, Grem JL. Phase I trial of concurrent stereotactic body radiotherapy and nelfinavir for locally advanced borderline or unresectable pancreatic adenocarcinoma. Radiother Oncol. 2019 Mar;132:55-62. doi: 10.1016/j.radonc.2018.11.002. Epub 2018 Dec 20. PMID 30825970